CLINICAL TRIAL: NCT05882344
Title: Cholinergic Deep Brain Stimulation for Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Christos Constantinidis, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240675
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease, Early Onset; Dementia; Alzheimer Disease
Keywords: Stimulation; Nucleus Basalis; Alzheimer; Memory
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: This is a feasibility study to investigate the potential of Deep Brain Stimulation to improve cognitive abilities and counteract the effects of Alzheimer's disease. Deep Brain Stimulation electrodes targeting the Nucleus Basalis of Meynert (NB) will be implanted bilaterally in patients. NB is the sole source of acetylcholine to the neocortex. Such stimulation may not only treat the cognitive symptoms but may have disease-modifying effects. Intermittent stimulation will be delivered at 60 pulses per second for 20 seconds of each minute for one hour per day. The study design will test the safety and feasibility of stimulation, potential benefits in cognitive function assessed with a battery of neurocognitive tests, cholinergic neurotransmission evaluated with Positron Emission Tomography, and ability to reverse Alzheimer's biomarkers, including beta amyloid and tau in the cerebrospinal fluid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Patients who are implanted and receive intermittent stimulation daily for the first 12 months
  Interventions: Procedure: Device Implantation- Boston Scientific, VERCISE GENUS™ system; Device: DBS Stimulation - Boston Scientific, VERCISE GENUS™ system

INTERVENTIONS:
Procedure: Device Implantation- Boston Scientific, VERCISE GENUS™ system — Participants will be implanted with DBS leads bilaterally, targeting the Nucleus Basalis of Meynert. The study team will record Local Field Potentials with and without stimulation, intraoperatively. These results will help the team determine at the end of the study whether LFP desynchronization (decrease in 5-15 Hz power), or other physiological signature, can be used to predict the location that provides the most effective intervention. Finally, the team will also ascertain the safety of the procedure and NB stimulation itself.
Device: DBS Stimulation - Boston Scientific, VERCISE GENUS™ system — Daily intermittent stimulation (60 Hz x 20s/min)

SUMMARY:
This project will investigate the potential of Deep Brain Stimulation to improve cognitive abilities and counteract the effects of Alzheimer's disease. Deep Brain Stimulation electrodes targeting the Nucleus Basalis of Meynert (NB) will be implanted bilaterally in a cohort of patients. NB is the sole source of acetylcholine to the neocortex. Such stimulation may not only treat the cognitive symptoms but may have disease-modifying effects. Drawing from animal experiments in non-human primates that showed success of this approach, intermittent stimulation will be delivered at 60 pulses per second for 20 seconds of each minute for one hour per day. The study team will recruit patients, shortly after first being diagnosed with Alzheimer's disease. The study design will test the safety and efficacy of stimulation, potential benefits in cognitive function assessed with a battery of neurocognitive tests, cholinergic neurotransmission evaluated with Positron Emission Tomography, and ability to reverse Alzheimer's biomarkers, including beta amyloid and tau in the cerebrospinal fluid. Successful completion of this project will lead to a potential new intervention for the cognitive impairments of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Probable, early-stage AD, as defined by NIA-AA 2018 criteria, including amnestic Mild Cognitive Impairment (MCI)

  * Clinical Dementia Rating (CDR) global score of 0.5-1.0 with a memory box score of at least 0.5
  * MMSE ³ 23
  * Stable cognitive enhancer medication equivalent to 10 mg/day donepezil or less for at least 60 days
  * Stable other medications (e.g., psychotropics)
  * Valid informed consent if female, subjects who are post-menopausal or surgically sterile or willing to use birth control methods for the duration of the study
  * an available caregiver willing to participate
  * subject is living at home and likely to remain at home for the study duration.

Exclusion Criteria:

* Active or unstable psychiatric illness
* Inability to tolerate general anesthesia.
* Another concurrent CNS condition or clinical co-morbidity interfering with the study (ie, stroke, Parkinson's disease, Lewy-Body dementia or other form of dementia, other evidence of significant structural brain pathology).
* Current major psychiatric disorder such as schizophrenia, bipolar disorder or major depressive disorder based on psychiatric consult at screening visit
* Verbal IQ<85
* Contraindication regarding anesthesia, stereotactic operation, MRI (e.g. claustrophobia, or implants), or PET (e.g. insulin dependent diabetes) procedures
* Inability to undergo PET or MRI imaging
* Active alcohol or substance abuse as defined by DSM5
* Is unable or unwilling to comply with protocol follow-up requirements
* Is actively enrolled in another concurrent clinical trial.
* Terminal illness associated with expected survival of <12 months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating score change | 12 - 24 Months
  . The primary outcome indicating success will be an increase in the mean score of the Clinical Dementia Rating - Sum of Boxes of the pre-stimulation baseline that is equal or greater than the increase in the post-stimulation data by 1 point or more, after 12-36 months of stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Blake, PhD, Principal Investigator — Augusta University; Dario Englot, MS, PhD, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
This experiment will generate behavioral/cognitive assessment, imaging data, and biochemical assays under intermittent stimulation of the nucleus basalis from 2 patients. De-identified, quality-controlled raw data sets and documentation for the processed data will be made available for research purposes, in accordance with Vanderbilt IRB policy for sharing de-identified data to maximize dissemination. All data will be de-identified prior to receipt by the repository, but the information needed to generate a unique identifier (Digital Object Identifier [DOI]) will be collected for each subject. Data will be archived and shared using the Open Science Framework (OSF) repository, which is a widely accessible, open, and secure online platform for sharing scientific data and documentation. Data analysis will be performed using MATLAB and Python; these scripts will be made available on our GitHub lab website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available at the time of an associated publication or at the end of the project period, whichever comes first. Unpublished data will also be made available at the end of the project period. Data will continue to be shared for a minimum of five years after the end of the project period.
Access Criteria: Data will be freely available at OSF, and any research can access the data by creating a free OSF account.

REFERENCES:
- [Background] Koh EJ, Golubovsky JL, Rammo R, Momin A, Walter B, Fernandez HH, Machado A, Nagel SJ. Estimating the Risk of Deep Brain Stimulation in the Modern Era: 2008 to 2020. Oper Neurosurg. 2021 Oct 13;21(5):277-290. doi: 10.1093/ons/opab261. PMID 34392372
- [Background] Kuhn J, Hardenacke K, Lenartz D, Gruendler T, Ullsperger M, Bartsch C, Mai JK, Zilles K, Bauer A, Matusch A, Schulz RJ, Noreik M, Buhrle CP, Maintz D, Woopen C, Haussermann P, Hellmich M, Klosterkotter J, Wiltfang J, Maarouf M, Freund HJ, Sturm V. Deep brain stimulation of the nucleus basalis of Meynert in Alzheimer's dementia. Mol Psychiatry. 2015 Mar;20(3):353-60. doi: 10.1038/mp.2014.32. Epub 2014 May 6. PMID 24798585
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Todd S, Barr S, Passmore AP. Cause of death in Alzheimer's disease: a cohort study. QJM. 2013 Aug;106(8):747-53. doi: 10.1093/qjmed/hct103. Epub 2013 May 7. PMID 23653484
- [Background] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413
- [Background] Williams MM, Storandt M, Roe CM, Morris JC. Progression of Alzheimer's disease as measured by Clinical Dementia Rating Sum of Boxes scores. Alzheimers Dement. 2013 Feb;9(1 Suppl):S39-44. doi: 10.1016/j.jalz.2012.01.005. Epub 2012 Aug 1. PMID 22858530